CLINICAL TRIAL: NCT00988130
Title: HIFU Lesion Control in Patients With Non-metastatic Progressive Prostate Cancer
Brief Title: High-Intensity Focused Ultrasound Focal Ablation in Treating Patients With Progressive Prostate Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University College London Hospitals (Other)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000652331; UCL-09-H0714-7; EU-20977
Record Dates: First submitted 2009-09-30; First posted 2009-10-01 (Estimated); Last update posted 2013-08-26 (Estimated); Status verified 2011-05

CONDITIONS: Prostate Cancer; Sexual Dysfunction
Keywords: sexual dysfunction; stage I prostate cancer; stage IIB prostate cancer; stage IIA prostate cancer; stage III prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms; Sexual Dysfunction, Physiological | interventions — High-Intensity Focused Ultrasound Ablation

INTERVENTIONS:
Other: laboratory biomarker analysis
Other: questionnaire administration
Procedure: assessment of therapy complications
Procedure: high-intensity focused ultrasound ablation
Procedure: quality-of-life assessment

SUMMARY:
RATIONALE: High-intensity focused ultrasound focal ablation uses high-energy sound waves to kill tumor cells.

PURPOSE: This phase II trial is studying the side effects of high-intensity focused ultrasound focal ablation and to see how well it works in treating patients with progressive prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To evaluate the side effects of high-intensity focused ultrasound (HIFU) ablation in men with non-metastatic progressive prostate cancer.
* To evaluate the quality of life of patients treated with this regimen.

Secondary

* To determine the success of index lesion ablation with HIFU at 6 months after treatment by demonstrating the absence of cancer in the treated or ablated area by transrectal ultrasound biopsy.
* To evaluate the prostate-specific antigen kinetics after index lesion ablation in patients treated with this regimen.
* To evaluate the proportion of men who require androgen blockade at 12 months of follow-up.

OUTLINE: Patients undergo focal ablation with high-intensity focused ultrasound (HIFU) ablation on day 1. Treatment may repeat at 6 months in patients with progressive disease.

Blood samples and prostate biopsies are collected periodically for further analysis.

Patients complete questionnaires (IPSS, IPSS-QoL, ICS, IIEF-5, and FACT-P) at baseline and periodically during study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed prostate cancer by transrectal or transperineal template prostate biopsies

  * Stage ≤ T3bN0M0
  * Gleason grade ≤ 8
  * Serum PSA ≤ 20 ng/mL
  * Bone scan- or cross-sectional imaging-negative for metastatic or nodal (outside prostate) disease
  * No metastatic disease and/or nodal spread by CT scan or MRI
* Index lesion or other secondary lesions with a volume ≥ 0.5 cc by MRI
* No prostatic calcification and cysts (on transrectal ultrasound) that would interfere with effective delivery of therapy

PATIENT CHARACTERISTICS:

* Able to tolerate a transrectal ultrasound
* Not allergic to latex
* Fit for major surgery as assessed by a consultant anaesthetist
* Able to have MRI scanning (i.e., none of the following conditions: severe claustrophobia, permanent cardiac pacemaker, metallic implant, etc.)

PRIOR CONCURRENT THERAPY:

* No prior radiotherapy
* No androgen suppression and/or hormone treatment within the past 12 months
* No prior significant rectal surgery preventing insertion of transrectal high-intensity focused ultrasound (HIFU) probe (decided on the type of surgery in individual cases)
* No prior transurethral resection of the prostate (or equivalent procedures) within the past 2 years
* No prior HIFU, cryosurgery, thermal, or microwave therapy to the prostate

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2009-07

PRIMARY OUTCOMES:
Total proportion of men with erectile dysfunction and/or incontinence
Quality of life

SECONDARY OUTCOMES:
Success of index lesion ablation with HIFU at 6 months
Prostate-specific antigen kinetics
Proportion of men requiring androgen blockade at 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Mark Emberton, MD, FRCS, MBBS, Principal Investigator — University College London Hospitals
Locations (1):
- University College Hospital - London, London, England, United Kingdom

REFERENCES:
- [Derived] Ahmed HU, Dickinson L, Charman S, Weir S, McCartan N, Hindley RG, Freeman A, Kirkham AP, Sahu M, Scott R, Allen C, Van der Meulen J, Emberton M. Focal Ablation Targeted to the Index Lesion in Multifocal Localised Prostate Cancer: a Prospective Development Study. Eur Urol. 2015 Dec;68(6):927-36. doi: 10.1016/j.eururo.2015.01.030. Epub 2015 Feb 11. PMID 25682339